CLINICAL TRIAL: NCT04149964
Title: Postoperative Pain Control in Septum and Sinus Surgery: A Novel Approach.
Brief Title: Postoperative Pain Control in Septum and Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, David Seel, Principal Investigator, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-259
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Results first posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Post-operative Pain; Sinus Surgery
Keywords: Post-operative pain; Sinus pain; Sinus surgery; Septum Pain; deviated septum
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Tablets; Oxycodone; Aspirin-oxycodone hydrochloride-oxycodone terephthalate combination; oxycodone-acetaminophen; Hydrocodone

STUDY DESIGN:
Intervention Model Description: Open, randomized into one of two arms study. Study arm 1: Standard of care arm of Acetaminophen (Tylenol) 325 mg every 6 hours as needed plus acetaminophen/hydrocodone 7.5 mg/325mg every 4 hours for breakthrough pain. Study arm 2: Acetaminophen 650 mg. every 6 hours round the clock plus 5 mg oxycodone every 4 hours as needed for breakthrough pain.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care arm (Active Comparator): Standard of Care Post-operative pain medication, Acetaminophen 325 mg every 6 hours as needed for pain plus acetaminophen/hydrocodone 7.5 mg/325 mg 1 tab every 4 hours as needed for pain.
  Interventions: Drug: Acetaminophen 325 mg Oral Tablet; Drug: Acetaminophen/Hydrocodone 325 mg/7.5 mg oral tablet
- Study Arm (Experimental): Acetaminophen 650 mg 1 tab every 6 hours round the clock plus Oxycodone 5 mg 1 tab every 6 hours as needed for breakthrough pain,.
  Interventions: Drug: Acetaminophen 650 mg Oral Tablet; Drug: OxyCODONE 5 mg Oral Tablet

INTERVENTIONS:
Drug: Acetaminophen 325 mg Oral Tablet — Standard of Care Acetaminophen 325 mg every 6 hours as needed for pain
  Other Names: Tylenol Standard Strength
  Arms: Standard of Care arm
Drug: Acetaminophen 650 mg Oral Tablet — Acetaminophen 650 mg scheduled every 6 hours round the clock for pain
  Other Names: Tylenol Extra Strength
  Arms: Study Arm
Drug: OxyCODONE 5 mg Oral Tablet — Oxycodone 5 mg every 4 hours as needed for breakthrough pain
  Other Names: Percodan, Percocet
  Arms: Study Arm
Drug: Acetaminophen/Hydrocodone 325 mg/7.5 mg oral tablet — Acetaminophen 325 mg/ Hydrocodone 7.5 mg oral tablet every 4 hours as needed for breakthrough pain
  Other Names: Norco
  Arms: Standard of Care arm

SUMMARY:
This study will evaluate if the use of acetaminophen round the clock (scheduled doses) will lead to less opiate use in the first week post-operative (after surgery) in sinus/septum surgery patients. Participants will be randomized like a flip of a coin to either the standard of care pain treatment of acetaminophen 325 mg as needed for pain plus opiates (acetaminophen/hydrocodone) as needed for breakthrough pain; OR to the study arm of acetaminophen 650 mg every 6 hours plus opiates (Oxycodone)as needed for breakthrough pain.

DETAILED DESCRIPTION:
Pain control in the postoperative period following septum and/or sinus surgery is controversial, as there is no consensus statement regarding current guidelines to direct clinical practice. Recent legislation limits opioid prescription length to 5 days only, which brings into question whether legislation will affect prescribing practices of physicians and whether or not giving patients an alternative to opiates will be a more efficacious route.

Current prescribing practices for septum and sinus surgery of the Otolaryngology private practice group includes as-needed acetaminophen 325 mg and as-needed acetaminophen/hydrocodone 7.5 mg/325 mg. If it can be demonstrated that use of 650 mg acetaminophen in scheduled doses of every 6 hours can decrease postoperative opiate use in the first week without significantly increase in patient pain, this may be deployed as an effective strategy of pain control as the use of opiates has come under scrutiny and attempts are being made to decrease or limit the use of these medications in the medical setting.

This study would look to demonstrate that scheduled doses of acetaminophen as opposed to reactionary as-needed acetaminophen can control post-operative pain to the point where narcotics would not be necessary.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing primary sinus surgery, primary septum surgery, or primary sinus/septum surgery
* 18 years of age or older
* Male or female
* No known allergies to or contraindications to the use of acetaminophen, hydrocodone, or oxycodone
* Patients discharged to home after surgery

Exclusion Criteria:

* Undergoing revision sinus, septum, or sinus/septum surgery
* Younger than 18 years old
* Allergy or contraindication to acetaminophen, hydrocodone, or oxycodone
* Patients admitted to the hospital postoperatively for airway monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Seel, DO., Principal Investigator — William Beaumont Hospital - Farmington Hills
Locations (1):
- Beaumont Hospital, Farmington Hills, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care Arm | Study Arm
Started | 34 | 31
Completed | 15 | 13
Not Completed | 19 | 18
Not completed — Lost to Follow-up | 19 | 18

BASELINE CHARACTERISTICS:
Population: 65 patients were enrolled. Baseline data on sex is not available for patients lost to follow up who did not complete post-operative questionnaire. 19 patients in SOC arm and 18 in study arm were lost to follow up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Arm | Study Arm | Total
Number analyzed (Participants) | 34 | 31 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.73 (15.40) | 46 (14.26) | 44.34 (6.79)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 65 patients were enrolled. Baseline data on sex is not available for patients lost to follow up who did not complete post-operative questionnaire. 19 patients in SOC arm and 18 in study arm were lost to follow up.
  Participants
    number analyzed (Participants) | 15 | 13 | 28
    Female | 10 | 4 | 14
    Male | 5 | 9 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 34 | 31 | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Doses of Opiate (Narcotic) Pain Medication
Description: Number of doses of opiates (narcotic) pain medication participants took for breakthrough pain in the first postoperative week.
Time Frame: 7 days
Population: 65 patients were enrolled. Data is not available for patients lost to follow up who did not complete post-operative questionnaire. 19 patients in SOC arm and 18 in study arm were lost to follow up.
Measure: Median (Inter-Quartile Range); unit: number of doses
Arm/Group | Standard of Care Arm | Study Arm
Number analyzed (Participants) | 15 | 13
number of doses | 1.0 [0 to 4.5] | 1.5 [0 to 6]

2. Secondary Outcome: Highest Subjective Pain Score
Description: Highest post-operative pain score during the first postoperative week as measured on an 11-point numeric pain scale from 0-10, with 0 = no pain and 10 = worst pain possible.
Time Frame: 7 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard of Care Arm | Study Arm
Number analyzed (Participants) | 15 | 13
score on a scale | 6.0 [4.25 to 7.0] | 5.0 [3.0 to 7.0]

3. Secondary Outcome: Lowest Subjective Pain Score
Description: Lowest post-operative pain score during the first postoperative week as measured on an 11 point numeric pain scale from 0-10, with 0 = no pain and 10 = worst pain possible.
Time Frame: 7 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard of Care Arm | Study Arm
Number analyzed (Participants) | 15 | 13
score on a scale | 2.0 [0.0 to 3.0] | 2.0 [0.0 to 2.0]

4. Secondary Outcome: Percentage of Time Participant Experienced Severe Pain
Description: Percentage of time participant experienced severe pain requiring breakthrough pain medication during the first postoperative week, as measured on an 11 point numeric scale, from 0% to 100%, where 0% means never in severe pain and 100% means always in severe pain.
Time Frame: 7 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Standard of Care Arm | Study Arm
Number analyzed (Participants) | 15 | 13
percentage of time | 0 [0 to 45] | 0 [0 to 30]

5. Secondary Outcome: Participant Use of Acetaminophen as Needed
Description: Number of participants who took acetaminophen as needed during the first postoperative week.
Time Frame: 7 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Study Arm
Number analyzed (Participants) | 15 | 13
Participants | 12 | 2

6. Secondary Outcome: Participant Use of Scheduled Acetaminophen Around the Clock
Description: Number of participants who took acetaminophen every 6 hours around the clock during first postoperative week.
Time Frame: 7 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Study Arm
Number analyzed (Participants) | 15 | 13
Participants | 3 | 11

7. Secondary Outcome: Chronic Use of Pain Medication
Description: Number of participants who answered "Yes" to the survey question, "Do you take pain medication, including narcotics, for any other medical condition?"
Time Frame: 7 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Study Arm
Number analyzed (Participants) | 15 | 13
Participants | 4 | 2

8. Secondary Outcome: Participant Use of Additional Pain Medication
Description: Number of participants who took other pain medication (over-the-counter or narcotic) in addition to study-prescribed pain medications during first postoperative week.
Time Frame: 7 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Study Arm
Number analyzed (Participants) | 15 | 13
Participants | 3 | 1

9. Secondary Outcome: Types of Other Pain Medication Used
Description: Self-reported name of pain medication (over-the-counter or narcotic) used by participants in addition to study-prescribed pain medications during the first postoperative week
Time Frame: 7 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Study Arm
Number analyzed (Participants) | 15 | 13
Participants
  Acetaminophen 325mg with 60mg codeine | 1 | 0
  morphine 15mg twice daily, 25mcg fentanyl | 0 | 1
  ibuprofen | 1 | 0
  None | 13 | 12

ADVERSE EVENTS:
Time Frame: 7 days
Description: 65 patients were enrolled. Data on adverse events including mortality is not available for patients lost to follow up who did not complete post-operative questionnaire. 19 patients in SOC arm and 18 in study arm were lost to follow up.
Arm/Group | Standard of Care Arm | Study Arm
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/15 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/64/NCT04149964/Prot_SAP_000.pdf